CLINICAL TRIAL: NCT04200742
Title: The Influences of Standardized Procedure of Bronchoalveolar Lavage on the Diagnosis of Pneumonia Pathogen of Critical Patients
Brief Title: Standardized BAL Procedure for Critical Patients to Diagnose Pneumonia Pathogens
Acronym: STABAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wu Jianfeng (Other)
Responsible Party: Sponsor-Investigator, Wu Jianfeng, chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: Standard BAL
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Bronchoalveolar Lavage; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, which is sampled by bronchoalveolar lavage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to improve the accuracy of the diagnosis of pulmonary pathogens and reduce the adverse impact of excessive BAL volume on patients, this study intends to explore the most optimal lavage volume in the middle lobe and the lower lobe of critical patients as well as seeking for the best way to manage BALF samples by means of detecting alveolar proteins and bacterial composition in BALF samples. The hypothesis is that the optimal lavage volume in the middle lobe and the lower lobe might be different. And to sample BALF separately through sequential lavage might be a better way to improve the accuracy of the diagnosis of pneumonia pathogens.

DETAILED DESCRIPTION:
This is a self-control study consisted of three parts. Firstly, searching for the optimal lavage volume in the middle lobe and the lower lobe of critical patients by exploring the differences between the concentration of alveolar proteins among BALF samples of every participant. Several BALF samples are seperately collected from every single participant through sequential lavage(an initial 20 ml saline lavage at main bronchus and 5 aliquots of 20 ml saline lavage at the subsegment of the right middle lobe or 6 aliquots of 20 ml saline lavage at the lower lobe) . The concentration of Alveolar proteins including Surfactant protein B (SP-B), Surfactant protein D (SP-D) and Human typeⅠprotein (HTⅠ-56) will be determined by enzyme-linked immunosorbent assay (ELISA). Meanwhile, the amount of living cells as well as the proportion of squamous cells and columnar cells in BALF samples will be counted. Secondly, to confirm the optimal lavage volume through quantitative bacterial culture of BALF and sputum samples of participants. And BALF samples will also be tested by next generation sequencing（NGS） to identify microorganism. Thirdly, to observe the effect of BAL on respiratory and cardiovascular systems. The Vital signs, arterial gas analysis, ventilator parameters and respiratory mechanical parameters of patients before and within 24 hours after the BAL procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit
* Mechanically ventilated patient
* 18 years old or above
* Pneumonia diagnosed by one of 1 - 4 plus 5

  1. purulent endotracheal secretions or increasing oxygen requirements;
  2. body temperature exceeds 38.0 ℃;
  3. potentially pathogenic bacteria be isolated from the endotracheal secretions;
  4. leukocyte count exceeds 10×10^9 per liter or less than 4×10^9 per liter;
  5. new or persistent radiographic features of pneumonia without another obvious cause.

Exclusion Criteria:

* considered to be unsuitable for bronchoscopy by attending physician;
* underwent bronchoalveolar lavage within the last 48 hours;
* medical history of lobectomy
* airway bleeding or pulmonary edema
* refuse to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is selected from the Departement of Critical Care Medicine of the First Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The optimal lavage volume at the middle lobe and the lower lobe, evaluated by the detection of SP-B, SP-D and HTⅠ-56 in bronchoalveolar lavage fluid (BALF). | 48 hours
  For the reason that SP-B, SP-D and HTⅠ-56 only exists in terminal airway and alveolus, the concentrations of them in BALF indicates the abundance of terminal airway materials obtained by bronchoalveolar lavage. SP-B, SP-D and HTⅠ-56 will be detected by enzyme-linked immunosorbent assay (ELISA).
The best way to manage BALF samples, evaluated by comparing the bacterial diversity and abundance in separately collected BALF specimens and mixed BALF specimen. | 3 days
  Mixed BALF specimen was a mixture of one tenth of separately collected BALF specimens. The BALF specimens will be cultured at 37℃，5% carbon dioxide for 18 to 24 hours, using blood ager, chocolate ager and MacConkey ager. Bacterial species will be identified by matrix-assisted laser desorption ionization-time of flight mass spectrometry (MALDI-TOF MS) and the colony counts will be recorded. Besides, BALF specimens will also be dectected by Next Generation Sequencing for the bacterial diversity and abundance. As a reference, culture of the endotracheal aspiration will be conducted.

SECONDARY OUTCOMES:
Quality of BALF samples, evaluated by counts of different kind of cells in BALF | 24 hours
  The living cells of BALF will be counted by Trypan blue staining. And the proportion of squamous cell and columnar cell will be counted by Wright-Giemsa staining.
Recovery of bronchoalveolar lavage fluid | 1 hour
  To record the volume of bronchoalveolar lavage fluid (BALF) recovered and calculate the recovery.
Impact of bronchoalveolar lavage (BAL) on the cardiovascular system. | 30 minutes before BAL; 15 minutes, 1 hours, 3 hours, 9 hours, 19 hours and 24 hours after BAL
  To observe the systolic arterial blood pressure (SAP), diastolic arterial blood pressure (DAP), mean arterial pressure (MAP) and heart rate (HR).
Change of pulmonary static compliance (Cst). | 30 minutes before BAL; 15 minutes, 1 hours, 3 hours, 9 hours and 24 hours after BAL.
  Cst will be measured with mechanical ventilator (Drager EvitaXL, Germany).
Chang of airway resistance (Raw). | 30 minutes before BAL; 15 minutes, 1 hours, 3 hours, 9 hours and 24 hours after BAL.
  Raw will be measured with mechanical ventilator (Drager EvitaXL, Germany).
Change of PaO2/FiO2 ratio. | About 2 hours before BAL; 15 minutes, 3 hours, 9 hours, 19 hours and 24 hours after BAL.
  PaO2 denotes the arterial oxygen partial pressure and FiO2 denotes the fraction of inspired oxygen.
Change of arterial carbon dioxide partial pressure (PaCO2). | About 2 hours before BAL; 15 minutes, 3 hours, 9 hours, 19 hours and 24 hours after BAL.
  PaCO2 will be measured by arterial blood gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Wu, M.D, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China